CLINICAL TRIAL: NCT06545981
Title: Ocular Perfusion in Patients With Idiopathic Intracranial Hypertension
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. Doz. Dr. med. univ., Medical University of Vienna
Other Study IDs: OPHT-241123
Record Dates: First submitted 2024-06-12; First posted 2024-08-09 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic intracranial hypertension (Group 1): 24 subjects with idiopathic intracranial hypertension
  Interventions: Other: Lumbar puncture and administration of medication
- Healthy control subjects (Group 2): 24 age- and sex-matched control subjects

INTERVENTIONS:
Other: Lumbar puncture and administration of medication — Patients with idiopathic intracranial hypertension will receive lumbar puncture and will be given medication to reduce intracranial pressure by neurologists. The lumbar puncture and the administration of medication are not part of this study, patients would also receive these without participating in the study.
  Groups: Idiopathic intracranial hypertension (Group 1)

SUMMARY:
The proposed study aims to evaluate optic nerve head blood flow and microcirculation in patients with idiopathic intracranial hypertension. For this purpose, optic nerve head blood flow will be examined in patients with IIH before and after therapy and additionally compared with healthy age- and sex-matched control subjects. In addition, other parameters will be measured, in particular retinal blood flow, retinal oxygen saturation and retinal neurovascular coupling.

DETAILED DESCRIPTION:
Idiopathic intracranial hypertension (IIH) is a neuroophthalmological disease, characterized by an increased intracranial pressure (ICP) without an identifiable causative factor. If not properly treated and carefully monitored the disease can even lead to irreversible severe or complete loss of vision or severe irreversible visual field defects, respectively. Given this clinical urgency, precise diagnostic tools become essential for timely decision making.

Laser Speckle Flowgraphy (LSFG) is a non-invasive, in-vivo imaging method, which quantitatively estimates blood flow in the optic nerve head, the choroid, the retina and the iris. LSFG has a low procedural complexity, obtains precise and reproducible measurements and is therefore suitable to assess ocular perfusion.

The proposed study aims to evaluate optic nerve head blood flow and microcirculation in patients with idiopathic intracranial hypertension. For this purpose, optic nerve head blood flow will be examined in patients with IIH before and after therapy and additionally compared with healthy age- and sex-matched control subjects. In addition, other parameters will be measured, in particular retinal blood flow, retinal oxygen saturation and retinal neurovascular coupling.

ELIGIBILITY:
Inclusion criteria for patients with idiopathic intracranial hypertension

* Men and Women aged ≥ 18 years
* Signed informed consent
* Newly diagnosed idiopathic intracranial hypertension or relapse of idiopathic intracranial hypertension
* Non-Smokers

Inclusion criteria for healthy age- and sex-matched control subjects

* Men and Women aged ≥ 18 years
* Signed informed consent
* Normal ophthalmic findings, unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the medical history, unless the investigator considers an abnormality to be clinically irrelevant
* Non-Smokers

Exclusion criteria for patients with idiopathic intracranial hypertension and healthy age- and sex-matched control subjects:

* Blood donation in the three weeks preceding the study
* Symptoms of a clinically relevant illness in the three weeks preceding the study
* Ocular inflammation or infection within the last 3 months
* History or family history of epilepsy
* Diabetes mellitus type 1 or type 2
* History or known presence of other cerebral vascular diseases (e.g.: arteriovenous malformation, aneurysm, major artery stenosis or occlusion)
* History or known presence of intracranial infections (e.g.: meningitis)
* History or known presence of other neurological diseases (e.g.: brain tumor, hydrocephalus, degenerative diseases)
* Patients receiving corticosteroids or immunosuppressant therapy
* Pregnant or breast-feeding women
* Women of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 48 patients will be included in the study:
  * Group 1: 24 subjects with idiopathic intracranial hypertension
  * Group 2: 24 age- and sex-matched control subjects
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Optic nerve head blood flow | Before the start of the therapy and 6 months after the start of the therapy
  Change in optic nerve head blood flow in patients with idiopathic intracranial hypertension before and 6 months after therapy (LSFG).

SECONDARY OUTCOMES:
Neurovascular coupling | Before the start of the therapy and 6 months after the start of the therapy
  Change in neurovascular coupling in patients with idiopathic intracranial hypertension before and 6 months after therapy (Dynamic Vessel Analyzer, IMEDOS, Jena, Germany)
Retinal nerve fiber layer thickness | Before the start of the therapy and 6 months after the start of the therapy
  Change in retinal nerve fiber layer thickness in patients with idiopathic intracranial hypertension before and 6 months after therapy.
Retinal and retinal layer thickness | Before the start of the therapy and 6 months after the start of the therapy
  Change in retinal and retinal layer thickness in patients with idiopathic intracranial hypertension before and 6 months after therapy (OCT).
Retinal vessel density | Before the start of the therapy and 6 months after the start of the therapy
  Change in retinal vessel density in patients with idiopathic intracranial hypertension before and 6 months after therapy (OCT-A).
Choroidal vascularity index (EDI-OCT) | Before the start of the therapy and 6 months after the start of the therapy
  Change in choroidal vascularity index (CVI is defined as the ratio of vascular luminal area (LA) to total choroidal area (TCA) and is presented as a percentage) in patients with idiopathic intracranial hypertension before and 6 months after therapy (EDI-OCT).
Retinal vessel diameter | Before the start of the therapy and 6 months after the start of the therapy
  Change in retinal vessel diameter (µm) in patients with idiopathic intracranial hypertension before and 6 months after therapy (retinal oximetry).
Optic nerve head blood flow | Before the start of the therapy and 6 months after the start of the therapy
  Change in optic nerve head blood flow in patients with idiopathic intracranial hypertension before and 6 months after therapy (LDF).
Retinal oxygen extraction | Before the start of the therapy and 6 months after the start of the therapy
  Change in retinal oxygen extraction in patients with idiopathic intracranial hypertension before and 6 months after therapy (LSFG, retinal oximetry).
Ocular perfusion pressure and arterial blood pressure | Before the start of the therapy and 6 months after the start of the therapy
  Change in ocular perfusion pressure and arterial blood pressure in patients with idiopathic intracranial hypertension before and 6 months after therapy.
Retinal oxygen saturation | Before the start of the therapy and 6 months after the start of the therapy
  Retinal oxygen saturation (SO2) in patients with idiopathic intracranial hypertension before and 6 months after therapy (retinal oximetry).
Choroidal thickness (EDI-OCT) | Before the start of the therapy and 6 months after the start of the therapy
  Change in choroidal thickness (µm) in patients with idiopathic intracranial hypertension before and 6 months after therapy (EDI-OCT).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Markey KA, Mollan SP, Jensen RH, Sinclair AJ. Understanding idiopathic intracranial hypertension: mechanisms, management, and future directions. Lancet Neurol. 2016 Jan;15(1):78-91. doi: 10.1016/S1474-4422(15)00298-7. Epub 2015 Dec 8. PMID 26700907
- [Background] Pruckner P, Mitsch C, Macher S, Krajnc N, Marik W, Novak K, Wober C, Pemp B, Bsteh G. The Vienna idiopathic intracranial hypertension database-An Austrian registry. Wien Klin Wochenschr. 2024 Jan;136(1-2):32-39. doi: 10.1007/s00508-023-02252-x. Epub 2023 Aug 31. PMID 37650963
- [Background] Wang MTM, Bhatti MT, Danesh-Meyer HV. Idiopathic intracranial hypertension: Pathophysiology, diagnosis and management. J Clin Neurosci. 2022 Jan;95:172-179. doi: 10.1016/j.jocn.2021.11.029. Epub 2021 Dec 17. PMID 34929642
- [Background] Sugiyama T, Araie M, Riva CE, Schmetterer L, Orgul S. Use of laser speckle flowgraphy in ocular blood flow research. Acta Ophthalmol. 2010 Nov;88(7):723-9. doi: 10.1111/j.1755-3768.2009.01586.x. PMID 19725814
- [Background] Tamaki Y, Araie M, Tomita K, Nagahara M, Tomidokoro A, Fujii H. Real-time measurement of human optic nerve head and choroid circulation, using the laser speckle phenomenon. Jpn J Ophthalmol. 1997 Jan-Feb;41(1):49-54. doi: 10.1016/s0021-5155(96)00008-1. PMID 9147189
- [Background] Miller MM, Chang T, Keating R, Crouch E, Sable C. Blood flow velocities are reduced in the optic nerve of children with elevated intracranial pressure. J Child Neurol. 2009 Jan;24(1):30-5. doi: 10.1177/0883073808321050. PMID 19168816